CLINICAL TRIAL: NCT00251732
Title: Role of Pain Modulation in GERD Patients Who Failed Standard Dose PPI.
Brief Title: Role of Pain Modulation in GERD Patients Who Failed Standard Dose Proton Pump Inhibitors (PPI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Southern Arizona VA Health Care System (U.S. Federal Agency); Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Ronnie Fass MD, SArizonaVAHCS
Organization: Southern Arizona VA Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Merit Review Study
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: acid reflux studies; efficacy of PPI therapy; failing PPI therapy; GERD; Acid Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Antidepressive Agents; Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard dose (PPI) plus low dose TCA (Active Comparator): Standard dose Rabeprazole(PPI) plus low dose tricyclic antidepressant(TCA)
  Interventions: Drug: Standard dose (once daily) PPI plus low-dose antidepressant
- Double dose PPI (Active Comparator): Double dose proton pump inhibitor plus placebo
  Interventions: Drug: Double dose PPI plus evening placebo
- Standard dose PPI plus placebo x 2 (Placebo Comparator): Standard dose 20 mg. once daily plus Placebo before dinner and placebo before bedtime
  Interventions: Drug: Rabeprazole , placebo, placebo

INTERVENTIONS:
Drug: Standard dose (once daily) PPI plus low-dose antidepressant — 20 mg. rabeprazole plus low dose tricyclic antidepressant(TCA)
  Other Names: Aciphex-PPI; Nortriptyline-TCA
  Arms: Standard dose (PPI) plus low dose TCA
Drug: Double dose PPI plus evening placebo — 20 mg. twice daily with a placebo
  Other Names: Aciphex-PPI, rabeprazole
  Arms: Double dose PPI
Drug: Rabeprazole , placebo, placebo — 20 mg rabeprazole(PPI) once daily -a.m. placebo -p.m. placebo -bedtime
  Other Names: Aciphex-rabeprazole (PPI); Nortriptyline-low-dose tricyclic antidepressant (TCA)
  Arms: Standard dose PPI plus placebo x 2

SUMMARY:
The main objective of this study is to evaluate the role of pain modulation in GERD patients who fail to obtain clinical relief with standard dose (once daily) PPI. The study will compare the efficacy of 1) standard dose PPI plus low-dose tricyclic antidepressant (TCA) to, 2) double dose PPI to, 3) standard dose PPI and placebo to determine the relative symptom resolution and health related quality of life in GERD patients who fail standard dose PPI and are randomly assigned to one of these three groups.

DETAILED DESCRIPTION:
To evaluate the role of pain modulation in gastroesophageal reflux disease(GERD)patients who fail to obtain clinical relief with standard dose (once daily) proton pump inhibitor(PPI). The study will compare the efficacy; of 1)standard dose PPI plus low-dose tricyclic antidepressant (TCA) to, 2) double dose PPI to, 3) standard dose PPI and placebo to determine the relative symptom resolution and health related quality of life in GERD patients who fail standard dose PPI and are randomly assigned to one of these three groups.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Ages 18 to 75
* At least two episodes of heartburn per week while on PPI once daily
* Able to communicate with the investigator and comply with the requirements of the study
* Subjects who give written informed consent after being given a full description of the study.

Exclusion Criteria:

* Known allergy or intolerance to TCA
* Use of antidepressant or a diagnosis of depression
* History of serious arrhythmia or use of anti-arrhythmics
* History of seizures
* Subjects with significant co-morbidity, e.g., cardiovascular, respiratory, urogenital, renal, gastrointestinal, hepatic, hematologic, endocrine, neurologic or psychiatric.
* Evidence or history of drug abuse within the past 6 months
* Erosive esophagitis, esophageal ulceration, peptic stricture, Barret's esophagus, or adenocarcinoma of the esophagus on endoscopy.
* History of esophagogastric surgery
* Gastric or duodenal lesions (ulcer, tumor, etc)
* Women who are pregnant or of childbearing age who are not on contraception
* Patients who are unwilling or unable to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Symptom control after 6 weeks of treatment | 6 weeks
  To measure the outcome after 6 weeks of treatment

SECONDARY OUTCOMES:
Number of drop-outs due to poor symptom control | 6 weeks
  To measure the number of drop-outs due to poor symptom control.
Level of antacid consumption | 6 weeks
  To measure the level of antacid consumption due to poor symptom control.
Improvement in quality of life | 6 weeks
  To improve quality of life with GERD symptom control.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Fass, MD, Principal Investigator — SAVAHCS
Locations (1):
- Southern Arizona VA Health Care System, Tucson, Arizona, United States